CLINICAL TRIAL: NCT06970327
Title: Comparative Study on the Efficacy of Totally Laparoscopic Distal Gastrectomy and Pylorus-Preserving Gastrectomy for Early Gastric Cancer in the Middle Stomach
Brief Title: Totally Laparoscopic Distal Gastrectomy VS Pylorus-Preserving Gastrectomy for Early Gastric Cancer in the Middle Stomach
Status: Completed | Type: Observational
Sponsor: Changzhi Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: ChangzhiMC202307; Grant No. 2023MX009 (Other Grant/Funding Number: Shanxi Provincial Health Commission)
Record Dates: First submitted 2025-04-26; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TLPPG: Totally laparoscopic pylorus-preserving gastrectomy
- TLDG: Totally laparoscopic distal gastrectomy

SUMMARY:
With the development of laparoscopic technology, the surgical treatment of early gastric cancer (EGC) has shifted towards minimally invasive, precise, and function-preserving strategies. Totally laparoscopic distal gastrectomy (TLDG) and totally laparoscopic pylorus-preserving gastrectomy (TLPPG) are minimally invasive procedures. However, there is a lack of systematic evidence to directly compare their efficacies.

This study focuses on two fully laparoscopic techniques, TLDG and TLPPG, to address two key objectives: (1) whether TLPPG can avoid the long-term functional sequelae of TLDG while ensuring oncological safety, including complications (delayed gastric emptying, reflux, and dumping syndrome), postoperative quality of life (assessed via the PGSAS-37 scale), and survival outcomes; and (2) the balance between complications and survival in function-preserving surgery. The findings aim to provide critical technical parameters for individualized surgical decision-making in EGC.

DETAILED DESCRIPTION:
With the continuous advancement and innovation of laparoscopic technology, the surgical treatment paradigm for early gastric cancer (EGC) is undergoing a profound transformation, gradually evolving towards a more minimally invasive, precise, and function-preserving approach. In this context, Totally Laparoscopic Distal Gastrectomy (TLDG) and Totally Laparoscopic Pylorus-Preserving Gastrectomy (TLPPG) have emerged as two highly representative minimally invasive surgical procedures. Characterized by smaller incisions, reduced trauma, and relatively faster postoperative recovery, they have garnered extensive attention in the field of EGC treatment. However, despite their application in clinical practice, there is currently a lack of comprehensive and systematic evidence-based medical data that can directly and thoroughly compare their therapeutic effects.

This study will focus on these two advanced laparoscopic surgical techniques, TLDG and TLPPG, and conduct in-depth exploration around two core objectives. Firstly, it will evaluate whether TLPPG can effectively avoid the long-term functional sequelae potentially caused by TLDG while ensuring oncological safety. These sequelae include common complications such as delayed gastric emptying, reflux, and dumping syndrome. Additionally, the study will comprehensively assess patients' postoperative quality of life using the PGSAS-37 scale and further analyze the impact of the two surgical procedures on patients' survival outcomes. Secondly, it will delve into how to achieve the optimal balance between complication control and patients' survival benefits in function-preserving surgeries. Through rigorous data analysis and scientific demonstration, this study aims to provide crucial technical parameters and reliable decision-making bases for the formulation of personalized surgical plans for EGC patients, thereby promoting the development of minimally invasive treatment for early gastric cancer towards a more precise and efficient direction.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative diagnosis of early gastric adenocarcinoma (invasion limited to the mucosa or submucosa) confirmed by tissue biopsy, abdominal enhanced CT, and endoscopic ultrasound;
* Tumor located in the gastric body or distal stomach, >4 cm from the pylorus;
* Ineligible for endoscopic mucosal dissection or elected for surgical treatment by family;
* Complete clinical and pathological data.

Exclusion Criteria:

* Severe anemia, coagulation disorders, or gastric outlet obstruction;
* History of gastric or upper abdominal surgery;
* Concurrent malignant tumors, ascites, edema, or pleural effusion;
* Gastric ulcers, polyps, or intestinal metaplasia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 63 patients with TLDG and 32 with TLPPG were included. The two groups of patients had similar sex, age, body mass index (BMI), and preoperative hemoglobin and albumin levels.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Complications | From surgery completion to 30 days post - operation
  Incidence of postoperative complications classified by the Clavien-Dindo criteria, including rate of Infection, Anastomotic issues, and Delayed gastric emptying.

SECONDARY OUTCOMES:
Age | Baseline
  The age of the patient at the time of enrollment in the study.
Weight（Kilograms） | Baseline
  The weight of the patient.
Height（Centimeters） | Baseline
  The height of the patient.
Body Mass Index (BMI) | Baseline
  The body mass index of the patient, calculated as weight (kg) divided by height squared (m²).
Blood Loss（Milliliters） | Intraoperative
  The total volume of blood lost during the surgical procedure.
Operation Time（Minutes） | Intraoperative
  The total duration of the surgical procedure.
Number of Examined Lymph Nodes | Intraoperative
  The total number of lymph nodes examined during the surgical procedure.
Time to Flatus | Perioperative
  The time elapsed from the end of the surgery until the patient experiences the first flatus.
Time to Defecation | Perioperative
  The time elapsed from the end of the surgery until the patient has the first bowel movement.
Time to Bite & Sup | Perioperative
  The time elapsed from the end of the surgery until the patient is able to eat and drink normally.
Hospital Stay Duration | Perioperative
  The total number of days the patient remains hospitalized after the surgical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- HeJi hospital affiliated ChangZhi medical college, Changzhi, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided